CLINICAL TRIAL: NCT01196572
Title: Cold vs. Laser Internal Urethrotomy Treatment of Urethral Strictures
Brief Title: Efficiency of Cold vs. Laser Internal Urethrotomy Treatment of Urethral Strictures
Acronym: IU
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Dr. Barak Rosenzweig, Urology department, Sheba Hospital, Israel.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-10-7897-ZD-CTIL
Record Dates: First submitted 2010-09-04; First posted 2010-09-08 (Estimated); Last update posted 2011-08-09 (Estimated); Status verified 2011-08

CONDITIONS: Urethral Strictures
Keywords: stricture; urethra; laser; urethrotomy; holmium; bladder outlet obstruction
MeSH Terms: conditions — Urethral Stricture; Constriction, Pathologic; Urinary Bladder Neck Obstruction | interventions — Lasers, Solid-State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laser IU (Experimental): Urethral stricture incised by Holmium laser
  Interventions: Procedure: Internal Urethrotomy
- Cold knife IU (Active Comparator): Urethral stricture incised by knife
  Interventions: Procedure: Internal Urethrotomy

INTERVENTIONS:
Procedure: Internal Urethrotomy — surgical incision of urethral stricture using endoscopic cold knife vs. endoscopic laser
  Other Names: Holmium laser

SUMMARY:
The purpose of this study is to determine whether laser internal urethrotomy (IU) is as efficient as cold knife internal urethrotomy for treatment of anterior urethral strictures regarding post operative urination outflow, stricture recurrence rate and possible post- operative complications

DETAILED DESCRIPTION:
The current surgical treatment for anterior urethral stricture includes internal urethrotomy (IU) by cold knife. Recurrence rate after such procedure is quoted as 35-70% in 2 to 5 years follow-up. Possible surgical alternative procedures include: open surgical urethral re-construction, urethral stents usage & laser IU. According to existing data (Nd-YAG laser- retrospective) the recurrence rate after laser IU is far better comparing to cold knife urethrotomy. The current research intends to address this question using prospective randomized methods.

ELIGIBILITY:
Inclusion Criteria:

* Men over 18 years old with urethral stricture

Exclusion Criteria:

* S/P urethral reconstruction
* Posterior urethral strictures
* Children

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-09; Primary Completion 2012-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
post operative clinical & imaging signs of urinary outflow obstruction or partial obstruction | up to 2 years
  Urethral stricture & urinary flow will be assessed by physical examination, urethrography, cystoscopy, sonographic bladder scan for urine rest, urine flowmetry & clinical questionnaire (IPSS).

SECONDARY OUTCOMES:
post operative complications | up to 2 years
  Complications such as urinary tract infection (UTI), bladder outlet obstruction (BOO), catheter re-insertion & re-operations will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba_Medical_Center, Ramat Gan, Israel